CLINICAL TRIAL: NCT02160847
Title: Pilot Trial of the DRIVE Parent Training Curriculum to Target Risk Factors for Childhood Obesity
Brief Title: Development of the DRIVE Curriculum to Address Childhood Obesity Risk Factors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia State University (Other)
Collaborators: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Jenelle Shanley, Assistant Professor, Georgia State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5800752
Record Dates: First submitted 2014-06-06; First posted 2014-06-11 (Estimated); Results first posted 2018-10-26 (Actual); Last update posted 2018-12-17 (Actual); Status verified 2018-12

CONDITIONS: Pediatric Obesity
Keywords: children; pediatric obesity; parent training; home-based; nutrition; physical activity; parent-child interaction; parenting
MeSH Terms: conditions — Pediatric Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DRIVE program (Experimental): Participants in the experimental group will receive the DRIVE curriculum (15 sessions) via weekly sessions conducted in their home by a DRIVE provider.
  Interventions: Behavioral: DRIVE Program
- Control Group (No Intervention): The parents in the control group will be mailed information on nutrition, physical activity, and parent-child interactions. Information on nutrition will include guidelines provided by the "MyPlate" website (http://www.choosemyplate.gov/preschoolers.html) in addition to information on proper nutrition and suggest levels of physical activity for preschoolers. Lastly, parents will be provided with the free publication, "Adventures in Parenting: How responding, Preventing, Monitoring, Mentoring, and Modeling Can Help You Be A Successful Parent," authored by National Institutes of Health, Eunice Kennedy Shriver National Institute of Child Health and Human Development. Information covered in this document includes effective parenting strategies for children at specific ages.

INTERVENTIONS:
Behavioral: DRIVE Program — The DRIVE program (Developing Relationships that Include Values of Eating and Exercise) is a home-based parent training program, which involves 15 sessions focusing on parent-child interactions, health and nutrition, and physical activity
  Arms: DRIVE program

SUMMARY:
The purpose of this study is to help overweight or obese children to maintain or reduce their body mass index (BMI) through the home-based parent training program the investigators developed called DRIVE. The investigators hypothesize that children from families that receive the DRIVE program will show greater maintenance or improvement in their BMIs than families who do not receive DRIVE.

DETAILED DESCRIPTION:
The DRIVE program (Developing Relationships that Include Values of Eating and Exercise) is a home-based parent training program with 15 sessions focused on improve family nutrition and physical activity and promoting positive parent-child interactions. The aim of this study is to pilot-test the development of a childhood obesity program that includes parenting and health information. Participants in this study will be recruited through community organizations based upon their obesity health risk. Only families whose children's BMI percentile is greater than or equal to 75 will be eligible to participate in this study These participants will be randomly assigned to either the control group, in which participants will receive health information via mail only, or the experimental group that will participate in 15 DRIVE sessions focusing on parent-child interactions, health and nutrition, and physical activity. Both groups will complete a baseline assessment, mid-point assessment, and post assessment in their home, which will measure parent and child height, weight, and waist circumference; parent attitudes towards health and nutrition; and parent and child food consumption and physical activity levels. Results from this study will provide information regarding the feasibility of implementing the DRIVE curriculum as well as its impact on parent and child body mass indexes, and parents' knowledge, and attitudes related to nutrition.

ELIGIBILITY:
Inclusion Criteria:

* Child age 2-6 years old with a BMI percentile greater than or equal to 75
* Fluent in English
* Parent has primary custody of the primary child participant in the study

Exclusion Criteria:

* Pregnant or currently breastfeeding (parent)
* Planning to get pregnant while enrolled in the study (parent)
* Have BMI greater than 45 (parent)
* Chronic disease that affects body weight, appetite, or metabolism (for example, diabetes- type I or type II) (child)
* Have HIV or AIDS (child)
* Use prescription or over-the-counter medications or herbal products that affect appetite, body weight, or metabolism (child)
* Plan to move out of the Atlanta/Baton Rouge area for the duration of enrollment (approximately 5 months) (family)
* Plan to be out of the Atlanta/Baton Rouge area for more than 2 weeks for the duration of enrollment (approximately 5 months) (family)

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jenelle R Shanley, PhD, Principal Investigator — Georgia State University
Locations (2):
- United States (2):
  - Georgia State University, Atlanta, Georgia
  - Pennington Medical Center, Baton Rouge, Louisiana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barlow SE; Expert Committee. Expert committee recommendations regarding the prevention, assessment, and treatment of child and adolescent overweight and obesity: summary report. Pediatrics. 2007 Dec;120 Suppl 4:S164-92. doi: 10.1542/peds.2007-2329C. PMID 18055651
- [Background] Academy of Nutrition and Dietetics. Public Policy Priority Areas. n.d.; http://www.eatright.org/HealthProfessionals/content.aspx?id=7091#.URxVRGfAGnA.
- [Background] Centers for Disease Control and Prevention. Winnable Battles. n.d.; http://www.cdc.gov/WinnableBattles/index.html.
- [Background] Dietz WH, Gortmaker SL. Preventing obesity in children and adolescents. Annu Rev Public Health. 2001;22:337-53. doi: 10.1146/annurev.publhealth.22.1.337. PMID 11274525
- [Background] Han JC, Lawlor DA, Kimm SY. Childhood obesity. Lancet. 2010 May 15;375(9727):1737-48. doi: 10.1016/S0140-6736(10)60171-7. Epub 2010 May 5. PMID 20451244
- [Background] Haynos AF, O'Donohue WT. Universal childhood and adolescent obesity prevention programs: review and critical analysis. Clin Psychol Rev. 2012 Jul;32(5):383-99. doi: 10.1016/j.cpr.2011.09.006. Epub 2011 Sep 22. PMID 22681912
- [Background] Koplan JP, Liverman CT, Kraak VI; Committee on Prevention of Obesity in Children and Youth. Preventing childhood obesity: health in the balance: executive summary. J Am Diet Assoc. 2005 Jan;105(1):131-8. doi: 10.1016/j.jada.2004.11.023. No abstract available. PMID 15635359
- [Background] Ogden CL, Carroll MD, Kit BK, Flegal KM. Prevalence of obesity among adults: United States, 2011-2012. NCHS Data Brief. 2013 Oct;(131):1-8. PMID 24152742
- [Background] US Department of Health and Human Services. Strategic Plan for NIH Obesity Research: A Report of the NIH Obesity Research Task Force. 2011. http://obesityresearch.nih.gov/about/StrategicPlanforNIH_Obesity_Research_Full-Report_2011.pdf.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DRIVE Program | Control Group
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DRIVE Program | Control Group | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Child and parent population descriptions were separated for the demographic data.
  years
    Child: number analyzed (Participants) | 8 | 8 | 16
    Child | 3.88 (1.81) | 4.25 (1.67) | 4.06 (1.69)
    Parent: number analyzed (Participants) | 8 | 8 | 16
    Parent | 35.75 (5.04) | 34.5 (5.86) | 35.13 (5.32)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Child and parent population descriptions were separated for the demographic data.
  Participants
    Child: number analyzed (Participants) | 8 | 8 | 16
    Child: Female | 3 | 5 | 8
    Child: Male | 5 | 3 | 8
    Parent: number analyzed (Participants) | 8 | 8 | 16
    Parent: Female | 8 | 7 | 15
    Parent: Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Child and parent population descriptions were separated for the demographic data.
  Participants
    Child: number analyzed (Participants) | 8 | 8 | 16
    Child: Hispanic or Latino | 1 | 0 | 1
    Child: Not Hispanic or Latino | 7 | 8 | 15
    Child: Unknown or Not Reported | 0 | 0 | 0
    Parent: number analyzed (Participants) | 8 | 8 | 16
    Parent: Hispanic or Latino | 0 | 0 | 0
    Parent: Not Hispanic or Latino | 8 | 8 | 16
    Parent: Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Child and parent population descriptions were separated for the demographic data.
  Participants
    Child: number analyzed (Participants) | 8 | 8 | 16
    Child: American Indian or Alaska Native | 0 | 0 | 0
    Child: Asian | 0 | 0 | 0
    Child: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Child: Black or African American | 2 | 5 | 7
    Child: White | 5 | 3 | 8
    Child: More than one race | 1 | 0 | 1
    Child: Unknown or Not Reported | 0 | 0 | 0
    Parent: number analyzed (Participants) | 8 | 8 | 16
    Parent: American Indian or Alaska Native | 0 | 0 | 0
    Parent: Asian | 0 | 0 | 0
    Parent: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Parent: Black or African American | 2 | 5 | 7
    Parent: White | 6 | 3 | 9
    Parent: More than one race | 0 | 0 | 0
    Parent: Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Child BMIz
Description: The child's body mass index z-scores (BMIz) was calculated by dividing the the child's weight in kilograms (measured by a digital scale) by the child's height in meters (measured by a stadiometer). These measurements were taken at each assessment point (pre-, mid-, and post-assessment).
Time Frame: Week 0, Week 9, Week 19
Measure: Mean (Standard Deviation); unit: BMIz
Arm/Group | DRIVE Program | Control Group
Number analyzed (Participants) | 8 | 8
BMIz
  Change from Week 0 to Week 9 | -0.21 (0.53) | 0.26 (0.44)
  Change from Week 0 to Week 19 | -.05 (0.32) | 0.41 (.058)

2. Secondary Outcome: Change in Parent BMIz
Description: The parent's body mass index z-scores (BMIz) was calculated by dividing the the parent's weight in kilograms (measured by a digital scale) by the parent's height in meters (measured by a stadiometer). These measurements were taken at each assessment point (pre-, mid-, and post-assessment).
Time Frame: Week 0, Week 9, Week 19
Measure: Mean (Standard Deviation); unit: BMIz
Arm/Group | DRIVE Program | Control Group
Number analyzed (Participants) | 8 | 8
BMIz
  Change from Week 0 to Week 9 | -0.53 (0.83) | -0.69 (2.19)
  Change from Week 0 to Week 19 | -1.16 (1.44) | -0.59 (3.54)

ADVERSE EVENTS:
Time Frame: At each assessment point, Week 0, Week 9, and Week 19.
Arm/Group | DRIVE Program | Control Group
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes